CLINICAL TRIAL: NCT00462995
Title: Surgery for Early Lung Cancer With Preoperative Erlotinib (Tarceva): A Clinical Phase II Trial
Brief Title: Surgery for Early Lung Cancer With Preoperative Erlotinib (Tarceva): A Clinical Phase II Trial (SELECT)
Acronym: SELECT
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University Health Network, Toronto (Other)
Collaborators: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: UHN REB#: 06-0052-C
Record Dates: First submitted 2007-04-17; First posted 2007-04-19 (Estimated); Last update posted 2018-02-23 (Actual); Status verified 2018-02

CONDITIONS: Non Small Cell Lung Cancer
Keywords: Non Small Cell Lung Cancer; Lung Cancer; Erlotinib; Neoadjuvant Treatment
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung; Lung Neoplasms | interventions — Erlotinib Hydrochloride

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Erlotinib (Active Comparator): Erlotinib 150mg once a day p.o
  Interventions: Drug: Erlotinib

INTERVENTIONS:
Drug: Erlotinib — 150mg once a day for 28 days
  Other Names: Tarceva
Drug: Erlotinib — 28 days of Erlotinib before surgery in patients with stage I-IIb NSCLC

SUMMARY:
2.5 Rationale for preoperative erlotinib therapy

Erlotinib is the only EFGR tyrosine kinase inhibitor to demonstrate a survival advantage and symptom improvement in a large phase III trial after failure of chemotherapy in advanced non-small cell lung cancer (Shepherd, Rodrigues Pereira et al. 2005). Although the potential utility of erlotinib in earlier stage NSCLC is unclear, given its activity in advanced disease and its minimal toxicity profile, there is likely a subset of patients who may benefit and potentially be cured by adjuvant erlotinib therapy. Erlotinib may also have greater antitumour activity in earlier stage disease. Therefore, we propose a phase II study to assess erlotinib pre-operatively in clinical stage 1 and 2 NSCLC, and downstream effects on signal transduction pathways and possible markers of treatment resistance and sensitivity.

The proposed study involves administering oral erlotinib for four weeks (28 days) preoperatively in early stage (1A/B, 2A/B) NSCLC. Current waiting times for surgical resection of early stage NSCLC at UHN ranges from 4 to 6 weeks (Hui, Johnston et al. 2004), thus patients would not experience significant delay in time to surgery through this trial design. This study provides the opportunity to explore the impact of erlotinib on early stage NSCLC in humans, with pharmacodynamic assessment expected in 100% of patients post-treatment, in addition to correlative imaging. This study will evaluate the feasibility of preoperative therapy with erlotinib, and may facilitate the identification of predictive markers for response to erlotinib in early stage NSCLC. This may help further define the subset of patients who would benefit from adjuvant EGFR tyrosine kinase inhibitors, and those who may require other adjuvant approaches including chemotherapy and further clinical trials.

DETAILED DESCRIPTION:
Treatment will be administered on an outpatient basis. Patients may be identified by thoracic surgeons, respirologists and/or interventional chest radiologists for study participation upon clinical and radiographic assessment.

4.2 Diagnostic biopsy, Pretreatment Investigations

If patients have already had a core or FNA biopsy before referral, this material will be sought from the original pathologist for review and inclusion in the study with appropriate consent sought. If a patient does not have a biopsy upon presentation to the thoracic surgeon, and consents to inclusion in the trial, a percutaneous biopsy will be mandated as part of entry into the study. The order of test will be up to the treating thoracic surgeon. As part of this procedure a large localizing needle is inserted into the tumour. In collaboration with pathology, a fine needle is passed through the outer needle and an immediate diagnosis will be made at the time of fine needle aspiration biopsy. After a pathologic diagnosis of cancer is confirmed, additional biopsies to obtain material for correlative studies will be performed through the standard localizing needle, assuming no complications or technical difficulties have arisen. These studies will be done in collaboration with thoracic interventional radiologists from Diagnostic Imaging, who perform the lung fine needle aspirates and biopsies.

All patients will undergo pre-study assessments for symptoms, performance status, radiographic assessment and blood tests (complete blood count, electrolytes, liver and renal function tests). Blood samples before treatment and post treatment with erlotinib will be banked for future serum proteomic analysis. Assessment of response will occur after the 4-week treatment period. Toxicity will be assessed continuously, with patient assessment weekly on treatment, repeat blood tests at 2 weeks and imaging of measurable disease at 4 weeks. All subjects will be invited to have their initial diagnostic biopsy and subsequent surgical tumor specimen examined as part of the laboratory correlate component of the study. Patients will be considered evaluable for pharmacodynamic assessment if they complete at least 21 of the planned 28 days of therapy.

Patients will have PET-CT scan study done pre- and post-treatment (see section 7). If the enrolment PET-CT imaging reveals mediastinal disease (IIIA or IIIB) or extensive disease and this is pathologically confirmed the patient will not be enrolled in the study.

Once the diagnosis is established and assessment completed, oral erlotinib will be administered at a dose of 150 mg (1 pill) daily for 28 days prior to the planned mediastinoscopy and/or surgery. Tablets should be taken preferably in the morning with up to 200 mL of water at least 1 hour before or 2 hours after meals. If the patient forgets to take a dose, they should take the last missed dose as soon as they remember, as long as it is at least 12 hours before the next dose is due. If patient vomits after taking the dose, the dose may be retaken if the tablet is seen in the emesis. The last dose of erlotinib will be administered early in the morning of the mediastinoscopy or surgery.

If the mediastinoscopy reveals the presence of Stage III disease, the patient's mediastinoscopy samples may still be analyzed as part of the correlative study. Patients will be followed for 90 days or as long as required after the last dose of erlotinib to ensure resolution of any erlotinib-related toxicities. However these patients will be offered standard therapy for stage III disease off study protocol, for example a combination of chemotherapy, radiation with or without surgical resection. If these patients do proceed to thoracotomy post-chemotherapy and/or radiotherapy, their resection specimen will not be eligible for this correlative protocol.

ELIGIBILITY:
Inclusion Criteria:

* Patients must have cytology or biopsy-proven non-small cell lung carcinoma (NSCLC);
* Preoperative clinical stage must be 1A (T1N0), 1B(T2N0), 2A (T1N1) and 2B (T2N1) by radiographic criteria;
* Patients must be deemed appropriate candidates for resection by the treating surgeon and surgical assessment team;
* Patients must have measurable disease, defined as at least one lesion that can be accurately measured in at least one dimension (longest diameter to be recorded) as >20 mm with conventional techniques or as >10 mm with spiral CT scan;
* Age ³ 18 years;
* ECOG performance status £ 2 (Karnofsky ³ 60%; see Appendix A);
* Patients must have normal organ and marrow function as defined below:

  * absolute neutrophil count ³1,500/uL
  * platelets ³100,000/uL
  * total bilirubin £1.5 times institutional upper limit of normal
  * AST(SGOT)/ALT(SGPT) £2 times institutional upper limit of normal
  * creatinine £1.5 times institutional upper limit of normal , or creatinine clearance³50 mL/min/1.73 m2 for patients with creatinine levels above institutional normal;
* The effects of erlotinib on the developing human fetus are unknown. For this reason, women of childbearing potential and men must agree to use adequate contraception (abstinence, hormonal or barrier method of birth control) prior to study entry and for the duration of study participation. Should a woman become pregnant or suspect she is pregnant while participating in this study, she should inform her treating physician immediately;
* Patients on warfarin are not excluded from the trial but are required to have their INR measured intensively during the initial stages of starting the study drug as alterations in INR have been noted. This intensive monitoring should entail measurements (3 X week for the first week then twice weekly for the remainder of the trial);
* Ability to understand and the willingness to sign a written informed consent document

Exclusion Criteria:

* Patients clinically T2N1 (2B), and/or T3N0 (2B) requiring a sleeve lobectomy, and/or chest wall resection; and tumors with higher staging;
* Patients who have received prior anticancer treatment with chemotherapy, radiotherapy or EGFR inhibitor therapy;
* Patients who have had a previous diagnosis of cancer within 5 years are excluded except adequately treated non-melanoma skin cancer, and carcinoma in situ of the cervix or breast;
* Patients may not be receiving any other investigational or anticancer agents while on study;
* History of allergic reactions to erlotinib;
* Pre-existing diarrhea ³ NCI CTC Grade 2 (4 to 6 loose stools per day) not controlled on standard therapy;
* Uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, symptomatic congestive heart failure or evidence of cardiac dysfunction, unstable angina pectoris, cardiac arrhythmia, active peptic ulcer disease, poorly controlled diabetes mellitus, clinically significant or untreated ophthalmologic (e.g. Sjogrens etc.) or gastrointestinal conditions (e.g. Crohn's disease, ulcerative colitis) or psychiatric illness/social situations that would limit compliance with study requirements.
* Pregnant women are excluded from this study, as the effects of erlotinib on a developing fetus are unknown. Because there is an unknown but potential risk for adverse events in nursing infants secondary to treatment of the mother with erlotinib, breastfeeding should be discontinued if the mother is treated with this combination.
* HIV-positive patients receiving combination anti-retroviral therapy are excluded from the study because of possible pharmacokinetic interactions with erlotinib.
* Active malignancy at any other site including combined small cell and non-small cell carcinomas or a pulmonary carcinoid tumor;
* Because drugs that induce CYP3A4 enzymes have been shown to significantly reduce plasma concentrations of erlotinib, patients with ongoing use of phenytoin, rifampicin, carbamazepine, barbiturates, rifampicin, or St John's Wort are excluded;
* Incomplete healing from previous surgery;
* Use of any agent that decreases gastric pH, including proton pump inhibitors, histamine-2 receptor blockers or sodium bicarbonate. Use of calcium or magnesium based elixirs are not included;
* Concomitant use of CYP3A4 inhibitors, e.g. itraconazole, may result in increased levels of erlotinib (TARCEVA®). This increase may be clinically relevant since adverse experiences are related to dose and exposure.

Ages: 18 Years to 95 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2006-05; Primary Completion 2012-01 (Actual); Study Completion 2012-02 (Actual)

PRIMARY OUTCOMES:
changes in tumor cell proliferation measured by a 75% reduction of Ki67 Immunohistochemistry (ICH) expression comparing pre and postoperative lung cancer | Before surgery and after surgery

SECONDARY OUTCOMES:
response rate, stable disease rate evaluated by RECIST criteria, median overall and disease-free survival time, 1-year overall and disease-free survival rate, toxicity and time to disease progression | Baseline, 2weeks, 4weeks and 30 days after surgery

CONTACTS AND LOCATIONS:
Overall Officials: Natasha Leighl, MD FRCPC, Principal Investigator — University Health Network, Toronto; Thomas Waddell, MD FRCSC, Principal Investigator — University Health Network, Toronto
Locations (2):
- Canada (2):
  - Toronto General Hospital, Toronto, Ontario
  - Princess Margaret Hospital, Toronto, Ontario

REFERENCES:
- [Background] Shepherd, F. A., J. Pereira, et al. (2004).
- [Background] Parkin DM, Bray F, Ferlay J, Pisani P. Estimating the world cancer burden: Globocan 2000. Int J Cancer. 2001 Oct 15;94(2):153-6. doi: 10.1002/ijc.1440. No abstract available. PMID 11668491
- [Background] Pavelic K, Banjac Z, Pavelic J, Spaventi S. Evidence for a role of EGF receptor in the progression of human lung carcinoma. Anticancer Res. 1993 Jul-Aug;13(4):1133-7. PMID 8394672
- [Background] Soulieres D, Senzer NN, Vokes EE, Hidalgo M, Agarwala SS, Siu LL. Multicenter phase II study of erlotinib, an oral epidermal growth factor receptor tyrosine kinase inhibitor, in patients with recurrent or metastatic squamous cell cancer of the head and neck. J Clin Oncol. 2004 Jan 1;22(1):77-85. doi: 10.1200/JCO.2004.06.075. PMID 14701768
- [Background] Shepherd, F. A., J. Rodrigues Pereira, et al. (2005).
- [Background] Weber WA, Petersen V, Schmidt B, Tyndale-Hines L, Link T, Peschel C, Schwaiger M. Positron emission tomography in non-small-cell lung cancer: prediction of response to chemotherapy by quantitative assessment of glucose use. J Clin Oncol. 2003 Jul 15;21(14):2651-7. doi: 10.1200/JCO.2003.12.004. PMID 12860940
- [Background] Scagliotti GV, Selvaggi G, Novello S, Hirsch FR. The biology of epidermal growth factor receptor in lung cancer. Clin Cancer Res. 2004 Jun 15;10(12 Pt 2):4227s-4232s. doi: 10.1158/1078-0432.CCR-040007. PMID 15217963